CLINICAL TRIAL: NCT00237107
Title: Relation of Basal Cell Carcinoma Tumour Thickness, Histologically Estimated, in Punch Biopsies Performed Before and After Curretage.
Brief Title: Debulking Effect of Curretage on Basal Cell Carcinomas - a Histological Assessment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: EC-003
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Carcinoma, Basal Cell
Keywords: Cytoreduction Surgical Procedures; Curretage; Photochemotherapy
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- curettage (Experimental)
  Interventions: Procedure: Curretage

INTERVENTIONS:
Procedure: Curretage

SUMMARY:
The aim of this study was to compare histologically observed tumour infitration of basal cell carcinoma (bcc) lesions before and after curretage.A significant reduction of tumour depth would enable further bcc's included for superficial non-invasive treatment modalities such as topical photodynamic therapy.

ELIGIBILITY:
Inclusion Criteria:

* bcc with tumour depth two mm.or more

Exclusion Criteria:

* bcc tumours smaller than three mm in mean diameter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-04; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Reduction of tumour thickness 0,5mm or more after curretage | 1 hour

SECONDARY OUTCOMES:
Comparison of tumour thickness in punch biopsies performed on referral, before and after curretage. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eidi Christensen, MD, Principal Investigator — St. Olav University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Christensen E, Mork C, Foss OA. Pre-treatment deep curettage can significantly reduce tumour thickness in thick Basal cell carcinoma while maintaining a favourable cosmetic outcome when used in combination with topical photodynamic therapy. J Skin Cancer. 2011;2011:240340. doi: 10.1155/2011/240340. Epub 2011 Nov 15. PMID 22191035